CLINICAL TRIAL: NCT04102605
Title: Efficacy and Safety of Visual Perceptual Learning Using the Nunap Vision for Improvement of Visual Field Defect Caused by Brain Damage: Multi Center, Superiority Prove, Double-blind, Randomized, Confirmatory Study
Brief Title: Visual Perceptual Learning for the Treatment of Visual Field Defect
Acronym: VIVID2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nunaps Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DB_NV_P01
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Visual Fields Hemianopsia; Hemianopsia, Homonymous
Keywords: Visual field defect; visual perceptual learning; Humphrey visual field
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nunap Vision (Experimental): Nunap Vision , 5 days a week for 12 weeks
  Interventions: Device: Nunap Vision
- Nunap Vision-C (Sham Comparator): Nunap Vision-C, 5 days a week for 12 weeks
  Interventions: Device: Nunap Vision-C

INTERVENTIONS:
Device: Nunap Vision — Participants receive visual perceptual training using the Nunap Vision software
  Arms: Nunap Vision
Device: Nunap Vision-C — Participants receive sham training using the Nunap Vision-C software
  Arms: Nunap Vision-C

SUMMARY:
This study evaluates the efficacy of visual perceptual learning for the treatment of visual field defect caused by brain damage. Half of participants will receive visual perceptual training using the Nunap Vision, while the other half will receive sham training using the Nunap Vision-C.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years
* Brain damage-induced visual field defect
* At least 6 months after brain lesion
* Minimum of 4 testing locations, where measured threshold ≤ 20dB
* Verified visual pathway damage using CT or MRI
* K-MMSE(Korean Mini Mental Status Examination) score ≥ 24
* Visual acuity equal or better than 20/40
* Able to use the investigational device
* Patient/legally authorized representative has signed the informed consent form

Exclusion Criteria:

* Unreliable Humphrey visual field test (any of fixation loss, false positive, false negative ≥ 20%)
* Complete hemianopsia with sensitivity of the whole hemifield ≤ 3 dB
* Epilepsy, photosensitivity, Parkinson's disease
* Bilateral visual field defect
* Hemispatial neglect
* Ophthalmologic disorder that may interfere the trial
* Inability to discontinue psychostimulants such as methylphenidate, modafinil, and amphetamine.
* Candidate for carotid endarterectomy or stenting
* Received ophthalmologic surgery within 3 months, except for the cataract surgery
* Pregnant or breast feeding
* Participating in other clinical trial
* Any other condition that, in the opinion of the investigator, precludes participation in the trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Area of Humphrey visual field where sensitivity increased by equal or more than 6 dB relative to baseline | 12 weeks
  Improved regions have luminance sensitivity that increased by equal or more than 6 dB relative to baseline. The improved area ranges between 0 and 972 degree^2, of which larger area indicates better outcome.

SECONDARY OUTCOMES:
Changes in Humphrey visual field mean deviation relative to baseline | 12 weeks
  Changes in mean deviation value of whole field or defect field compared with the baseline value. The change of mean deviation ranges between -35 to +35 dB, of which higher value indicates better outcome.
Changes in scores of NEI-VFQ-25(the National Eye Institute Visual Function Questionnaire 25) relative to baseline | 12 weeks
  Changes in each components of NEI-VFQ-25 scores relative to baseline. The change of scores ranges between -100 to 100, of which higher value indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sun U. Kwon, MD, PhD, Study Chair — Asan Medical Center
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No